CLINICAL TRIAL: NCT05468112
Title: Improving Wellbeing of SHP Personnel at UAB
Acronym: SHPwell
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources for performance of project
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Keith McGregor, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008660
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stress, Psychological
Keywords: Mindfulness; Breathing; Meditation; Stress reduction; SKY Yoga
MeSH Terms: conditions — Stress, Psychological; Respiratory Aspiration | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This is a single group design in which participants participants are assigned to a SKY meditation treatment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sky Meditation and Mindfulness Intervention (Experimental): In person meditation classes will be 3 hours long on each of three consecutive days, and participants must be willing to attend all three sessions. An additional 7 online sessions will be delivered to participants in successive days after the initial in-person intervention. Participants will be asked to engage in daily 10 to 25 minute home resilience practice sessions performed five days per week. To support participants stabilization of the practices, optional daily guided practice will be offered online at a determined convenient time for all participants to allow full participation. The breathing techniques will be taught by certified instructors.
  Interventions: Behavioral: SKY Meditation and Mindfulness

INTERVENTIONS:
Behavioral: SKY Meditation and Mindfulness — The intervention is a 3-day in-person meditation and mindfulness workshop using the SKY meditation approach. It utilizes a unique set of standardized breathing techniques to rapidly reduce neuro-endocrine stress responses and the autonomic imbalance due to sympathetic overdrive, thus restoring autonomic homeostasis. These are interwoven with coping and stressor appraisal strategies, and simple stretching exercises. Classes will be 3 hours long on each of three consecutive days, and participants must be willing to attend all three sessions with an additional 7 consecutive days of online sessions immediately thereafter. In addition, participants will be asked to engage in daily 10 to 25 minute home resilience practice sessions performed five days per week. They will complete a follow-up session once per week in the subsequent 8 weeks.
  Other Names: SKY Yoga; Sudarshan Kriya Yoga

SUMMARY:
The main objective of this study is to evaluate the impact of a well-being program, SKY Campus Happiness, on well-being of students, faculties, and staff working/studying at School of Health Professional (SHP). SHP is leaning on the SKY Campus Happiness (SKY) program which is an integrative workshop format that includes both skill-building and group dynamics and may be critical for the effectiveness of the program. SKY is a university leadership and well-being program (campushappiness.org) that includes stress-management and tools for psychological resilience: yoga postures, breathing exercises, a breath-based meditation technique [Sudarshan Kriya Yoga]. SKY also includes positive psychology skills (e.g., gratitude, social connection, acts of kindness, meaning and purpose). In addition, the curriculum includes discussion and application of leadership skills and service learning. Relying on existing evidence of previous studies, we hypothesize that participating in this program will increase the well-being of people involved.

DETAILED DESCRIPTION:
Students/staff/faculties of SHP will be offered to participate in the SKY Breath Happiness workshop followed by participating in a research program designed to study the potential effectiveness of the SKY Breath Happiness Program as a stress-management, resilience building wellness tool in this population. They will be given an informed consent form to sign if they choose to participate in the study. The course that the students are enrolled in is the SKY program, which is an evidence-based bio-psycho-social program that utilizes a multi-dimensional relationship between biology and behavior. It utilizes a unique set of standardized breathing techniques to rapidly reduce neuro-endocrine stress responses and the autonomic imbalance due to sympathetic overdrive, thus restoring autonomic homeostasis. These are interwoven with coping and stressor appraisal strategies, and simple stretching exercises. Classes will be 3 hours long on each of three consecutive days, and participants must be willing to attend all three sessions. There will also be one mandatory one hour follow-up session one week later. Participants will be asked to engage in daily 10 to 25 minute home resilience practice sessions performed five days per week. To support participants stabilization of the practices, optional daily guided practice will be offered online at a determined convenient time for all participants to allow full participation. The breathing techniques will be taught by certified instructors.

ELIGIBILITY:
Inclusion criteria:

* Healthy students/faculty/staff who at UAB, School of Health Professionals
* Willingness to complete all study interventional components

Exclusion criteria:

* Inability to understand standard English
* Previous participation in a SKY intervention
* Pregnant persons
* Diagnosis of bipolar disorder or schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PERCEIVED STRESS SCALE | Pre/post-intervention with 8 week followup
  The Perceived Stress Scale(PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives.
Brief-COPE | Pre/post-intervention with 8 week followup
  The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.
Pittsburgh Sleep Quality Assessment | Pre/post-intervention with 8 week followup
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
Mini-Mood and Anxiety Symptom Questionnaire | Pre/post-intervention with 8 week followup
  The Mood and Anxiety Symptom Questionnaire (MASQ) is an instrument containing a range of symptoms relevant to depression and anxiety.
The Social Connectedness Scale - Revised | Pre/post-intervention with 8 week followup
  This scale assesses the degree to which persons feel connected to others in their social environment.
SF-12v2 | Pre/post-intervention with 8 week followup
  The SF-12v2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health.

SECONDARY OUTCOMES:
Open Ended Questions | Weekly after 8 weeks
  Qualitative questions of well-being
Focus Groups | After participation in sessions at 12 weeks
  Group discussion with transcript

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma A, Barrett MS, Cucchiara AJ, Gooneratne NS, Thase ME. A Breathing-Based Meditation Intervention for Patients With Major Depressive Disorder Following Inadequate Response to Antidepressants: A Randomized Pilot Study. J Clin Psychiatry. 2017 Jan;78(1):e59-e63. doi: 10.4088/JCP.16m10819. PMID 27898207
- [Background] Lai KSP, Watt C, Ionson E, Baruss I, Forchuk C, Sukhera J, Burhan AM, Vasudev A. Breath Regulation and yogic Exercise An online Therapy for calm and Happiness (BREATH) for frontline hospital and long-term care home staff managing the COVID-19 pandemic: A structured summary of a study protocol for a feasibility study for a randomised controlled trial. Trials. 2020 Jul 14;21(1):648. doi: 10.1186/s13063-020-04583-w. PMID 32665041
- [Result] Seppala EM, Bradley C, Moeller J, Harouni L, Nandamudi D, Brackett MA. Promoting Mental Health and Psychological Thriving in University Students: A Randomized Controlled Trial of Three Well-Being Interventions. Front Psychiatry. 2020 Jul 15;11:590. doi: 10.3389/fpsyt.2020.00590. eCollection 2020. PMID 32760296